CLINICAL TRIAL: NCT03335787
Title: The Long Term Effects Of Kinesio Taping On Balance In Patients With Stroke: A Single Blinded Randomized Controlled Trial
Brief Title: Effectiveness of Kinesio Taping On Balance In Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AbantIBU-Phys1
Record Dates: First submitted 2017-10-06; First posted 2017-11-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Athletic Tape; Proprioception; Hemiplegia; Gait
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Patients' information and contact will be obtained from neurologist and willing participant's gender, age and stroke onset data will be processed with a random number generator in order to form groups. Patients will divide into two groups as intervention and control with a normal distribution of gender, age and stroke onset.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both group will receive conventional stroke rehabilitation. Intervention group will receive Kinesio taping and control group would not receive a sham taping due to the possible sensory intervention of sham taping even though applying it without any stretch.
  Outcomes will be recorded by physical therapist using SPSS and groups would not be specified with letter. Statistical analysis will be conducted by another researcher who does not aware of groups given numbers on SPSS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Taping will be applied three times and will be reapplied one and two weeks later prior to first application for two weeks.
  Interventions: Other: Intervention
- Control (Other): Control group would not receive any taping in order to prevent sham taping sensory stimulation effect.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — Kinesio Tape apply to peroneal muscles in supine position starting from the peroneal muscle origin with using muscle activation technique by a certified KT1 and KT2 practitioner. Then ligament technique which will go through around ankle starting from medial and lateral metatarsophalangeal joints in order to improve ankle stability. Taping will be applied one week later and two weeks later prior to first application.
  Arms: Intervention
Other: Control — Any sham taping was not applied to the control group in order to prevent the sensory stimulant effect of taping. In order to achieve patients' blinding both groups participant will sign a same consent but control group will be called for taping a month later after study data collection completed.
  Arms: Control

SUMMARY:
The aim of this study is to investigate the long term effects of Kinesio taping applied on ankle and peroneal muscle in patients with stroke.

DETAILED DESCRIPTION:
Stroke is a common neurological problem and is one of the major causes of disability and death (1,2). In stroke patients, the mortality rate is approximately 30%, and there is an increase in the morbidity rate after stroke occurrence. In addition, stroke is one of the main factors in increases in the burden of health care expenses during adulthood (3).

There is a constant requirement for specific data about stroke rehabilitation methods for achieving evidence-based rehabilitation guidelines.To investigate the effects of repeated correction taping applied on the ankle and peroneus longus and peroneus brevis muscles on balance and gait in patients with stroke. Therefore, the aim of this study is to assess the long term effect of KT applied on ankle and peroneal muscle on both dynamic and static balance in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Diagnosed with Stroke
* Mini-Mental State Test score equal or above 25
* Modified Ashworth Scale Score lover then 3
* Able to walk 10 meter independently

Exclusion Criteria:

* Secondary neurological diseases
* Cognitive problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Balance evaluation systems test (BESTest)-Change from Baseline | two weeks
  BESTest contains 27 question under 6 subsections (biomechanical, stability limits, postural responses, anticipatory postural adjustments, sensory orientation, and dynamic balance during gait) all of which rates between 0 (unable) - 3 (normal function) points (22) was used to assess the dynamic and static balance during the activities. TUG was used to assess balance, mobility and walking ability of the patients before and after the procedure as a part of the BESTest. However, as a strong indicator of functional mobility we decided to analyze TUG results separately from the overall BESTest outcomes. Assessments will be conducted at baseline, after first application,one week later and 2 weeks later prior to first assessment.

SECONDARY OUTCOMES:
Functional reach test (FRT)-Change from Baseline | two weeks
  FRT was used to assess the limits of stability by measuring the distance that a patient can reach forward without losing balance. The test was performed while patient standing on both feet next to a wall. A measurement tape fixed to the wall on the level of patients' acromion. Cut of score was taken as 25 cm. Assessments will be conducted at baseline, after first application,one week later and 2 weeks later prior to first assessment.
Tetrax balance systems-Change from Baseline | two weeks
  Tetrax balance system which focuses measuring static balance and postural sways with integrated 4 force plates for tracking weight difference on forefoot and hindfoot. Primary principal of this device is to measure the center of mass and postural sways by using 4 force plates. Assessment was performed while patients standing on the force plates eyes facing forward and without touching anything with their hands. Normal values were taken as 1.0 standard deviation below and 1.5 standard deviation above the mean scores. Higher result related to somato-sensory dysfunction. For weight distribution index it is expected to %25 of total body weight recorded on each plate. Assessments will be conducted at baseline, after first application,one week later and 2 weeks later prior to first assessment.
Functional Independence Measure (FIM)-Change from Baseline | two weeks
  Index for measuring both motor and cognitive independency level of patients under total 18 questions. Scores vary from completely independent to completely dependent. Assessments will be conducted at baseline, after first application,one week later and 2 weeks later prior to first assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Çankaya, Ph.D, Study Director — Abant Izzet Baysal University; Ramazan Kurul, Ms.C, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After publication of article Tetrax balance scores, BESTest results and Timed Up and Go times can be shared with other researches with an excel data sheet. Researchers can contact corresponding researcher with his contact mail and request data.

REFERENCES:
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Wardlaw JM, Murray V, Berge E, del Zoppo GJ. Thrombolysis for acute ischaemic stroke. Cochrane Database Syst Rev. 2014 Jul 29;2014(7):CD000213. doi: 10.1002/14651858.CD000213.pub3. PMID 25072528
- [Background] Stroke Unit Trialists' Collaboration. Organised inpatient (stroke unit) care for stroke. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD000197. doi: 10.1002/14651858.CD000197.pub2. PMID 17943737
- [Background] Wade DT. Impact commentaries. Functional abilities after stroke: measurement, natural history and prognosis. J Neurol Neurosurg Psychiatry. 2012 Aug;83(8):770. doi: 10.1136/jnnp-2011-301689. Epub 2012 Jan 6. No abstract available. PMID 22228728
- [Background] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Background] Geiger RA, Allen JB, O'Keefe J, Hicks RR. Balance and mobility following stroke: effects of physical therapy interventions with and without biofeedback/forceplate training. Phys Ther. 2001 Apr;81(4):995-1005. PMID 11276182
- [Background] Geurts AC, de Haart M, van Nes IJ, Duysens J. A review of standing balance recovery from stroke. Gait Posture. 2005 Nov;22(3):267-81. doi: 10.1016/j.gaitpost.2004.10.002. Epub 2004 Dec 7. PMID 16214666
- [Background] Hillier S, Dunsford A. A pilot study of sensory retraining for the hemiparetic foot post-stroke. Int J Rehabil Res. 2006 Sep;29(3):237-42. doi: 10.1097/01.mrr.0000210052.32539.22. PMID 16900045
- [Background] de Haart M, Geurts AC, Huidekoper SC, Fasotti L, van Limbeek J. Recovery of standing balance in postacute stroke patients: a rehabilitation cohort study. Arch Phys Med Rehabil. 2004 Jun;85(6):886-95. doi: 10.1016/j.apmr.2003.05.012. PMID 15179641
- [Background] Mauritz KH. Gait training in hemiparetic stroke patients. Eura Medicophys. 2004 Sep;40(3):165-78. PMID 16172584
- [Background] Slupik A, Dwornik M, Bialoszewski D, Zych E. Effect of Kinesio Taping on bioelectrical activity of vastus medialis muscle. Preliminary report. Ortop Traumatol Rehabil. 2007 Nov-Dec;9(6):644-51. English, Polish. PMID 18227756
- [Background] Yoshida A, Kahanov L. The effect of kinesio taping on lower trunk range of motions. Res Sports Med. 2007 Apr-Jun;15(2):103-12. doi: 10.1080/15438620701405206. PMID 17578750
- [Background] Jaraczewska E, Long C. Kinesio taping in stroke: improving functional use of the upper extremity in hemiplegia. Top Stroke Rehabil. 2006 Summer;13(3):31-42. doi: 10.1310/33KA-XYE3-QWJB-WGT6. PMID 16987790
- [Background] Robbins S, Waked E, Rappel R. Ankle taping improves proprioception before and after exercise in young men. Br J Sports Med. 1995 Dec;29(4):242-7. doi: 10.1136/bjsm.29.4.242. PMID 8808537
- [Background] Fayson SD, Needle AR, Kaminski TW. The effects of ankle Kinesio taping on ankle stiffness and dynamic balance. Res Sports Med. 2013;21(3):204-16. doi: 10.1080/15438627.2013.792083. PMID 23777376
- [Background] Cortesi M, Cattaneo D, Jonsdottir J. Effect of kinesio taping on standing balance in subjects with multiple sclerosis: A pilot study\m1. NeuroRehabilitation. 2011;28(4):365-72. doi: 10.3233/NRE-2011-0665. PMID 21725170
- [Background] Yazici G, Guclu-Gunduz A, Bayraktar D, Aksoy S, Nazliel B, Kilinc M, Yildirim SA, Irkec C. Does correcting position and increasing sensorial input of the foot and ankle with Kinesio Taping improve balance in stroke patients? NeuroRehabilitation. 2015;36(3):345-53. doi: 10.3233/NRE-151223. PMID 26409338
- [Background] Palluel E, Nougier V, Olivier I. Do spike insoles enhance postural stability and plantar-surface cutaneous sensitivity in the elderly? Age (Dordr). 2008 Mar;30(1):53-61. doi: 10.1007/s11357-008-9047-2. Epub 2008 Mar 4. PMID 19424873
- [Background] Kilbreath SL, Perkins S, Crosbie J, McConnell J. Gluteal taping improves hip extension during stance phase of walking following stroke. Aust J Physiother. 2006;52(1):53-6. doi: 10.1016/s0004-9514(06)70062-9. PMID 16515423